CLINICAL TRIAL: NCT06615011
Title: Bardet Beidle Syndrome in a Syrian Adolescent : a Rare Case Report
Acronym: AlBaathU
Status: Not yet recruiting | Type: Observational
Sponsor: Al Baath University (Other)
Responsible Party: Principal Investigator, Shaghaf Alhallak, med student, Al Baath University
Other Study IDs: BBS syndrome
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Bardet Biedl Syndrome (BBS)
Keywords: Central obesity; Postaxial Polydactyly
MeSH Terms: conditions — Bardet-Biedl Syndrome; Obesity, Abdominal; Polydactyly, Postaxial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Bardet-Biedl Syndrome (BBS) is an uncommon genetic disorder that affects multiple organs. and presents with a variety of characteristics. It is caused by a dysfunction in the cilia. We present a case of bradet-biedl syndrome presenting with intellectual disabilities, post-axial polydactyly, gingival hyperplasia, and a significant family history of scleroderma. The diagnosis was determined based on clinical physical examination findings. The patient is undergoing treatment with Thyroxine. Although medical staff are incapable of treatment, systems support adjust the overall well-being and quality of life for individuals with Bardet-Biedl syndrome and their families.

DETAILED DESCRIPTION:
Bardet-Biedl Syndrome (BBS) is a rare genetic disorder that affects multiple organ systems presents with a variety of characteristics . It is caused by a dysfunction in the cilia The disorder is autosomal recessive and has a prevalence rate of 1 per 160000 live births in Europe. The primary manifestations include central obesity, post-axial polydactyly, retinal dystrophy, hypogonadism, learning difficulties, and renal malformations . Secondary manifestations include diabetes, brachydactyly, syndactyly, strabismus, cardiac problems, speech difficulties, and ataxia .The diagnosis of BBS requires the presence of four primary features or three primary features and two secondary features , a new paper suggests that modified criteria for diagnosis can be at a moderate level of confidence if it includes at least 2 primary criteria . In this paper, we describe an adolescent male with a unique presentation of BBS. To the best of our knowledge, this is the first case in Syria described in the literature

ELIGIBILITY:
Inclusion Criteria:

* any person

Exclusion Criteria:

* any person

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-12 (Estimated); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
bardet beidle syndrome | 2025

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ankleshwaria C, Prajapati B, Parmar S, Rathod V, Patel H, Dhorajiya D, Chavda N, Parmar K, Pathan F, Chauhan M. Bardet-Biedl Syndrome Presenting in Adulthood. Indian J Nephrol. 2022 Nov-Dec;32(6):633-636. doi: 10.4103/ijn.ijn_320_21. Epub 2022 Oct 2. PMID 36704599
- [Background] Oliaei F, Narimani H. Bardet-Biedl 9 Syndrome, A Rare Mutation. Iran J Kidney Dis. 2020 Mar;14(2):157-159. PMID 32165602
- [Background] Elawad OAMA, Dafallah MA, Ahmed MMM, Albashir AAD, Abdalla SMA, Yousif HHM, Daw Elbait AAE, Mohammed ME, Ali HIH, Ahmed MMM, Mohammed NFN, Osman FHM, Mohammed MAY, Abu Shama EAE. Bardet-Biedl syndrome: a case series. J Med Case Rep. 2022 Apr 29;16(1):169. doi: 10.1186/s13256-022-03396-6. PMID 35484558
- [Background] Dollfus H, Lilien MR, Maffei P, Verloes A, Muller J, Bacci GM, Cetiner M, van den Akker ELT, Grudzinska Pechhacker M, Testa F, Lacombe D, Stokman MF, Simonelli F, Gouronc A, Gavard A, van Haelst MM, Koenig J, Rossignol S, Bergmann C, Zacchia M, Leroy BP, Mosbah H, Van Eerde AM, Mekahli D, Servais A, Poitou C, Valverde D. Bardet-Biedl syndrome improved diagnosis criteria and management: Inter European Reference Networks consensus statement and recommendations. Eur J Hum Genet. 2024 Nov;32(11):1347-1360. doi: 10.1038/s41431-024-01634-7. Epub 2024 Jul 31. PMID 39085583
- [Background] Tsegaw A, Teshome T. Bardet-Biedl Syndrome in an Ethiopian. Int Med Case Rep J. 2021 Mar 19;14:177-181. doi: 10.2147/IMCRJ.S299421. eCollection 2021. PMID 33776488
- [Background] Shrinkhal, Singh A, Agrawal A, Mittal SK, Udenia H, Bandu GH. A rare case of Bardet-Biedl syndrome. Taiwan J Ophthalmol. 2019 Oct 17;10(2):138-140. doi: 10.4103/tjo.tjo_62_19. eCollection 2020 Apr-Jun. PMID 32874845